CLINICAL TRIAL: NCT01087372
Title: Stress Hyperglycemia in Critically Ill Patients. Potential Role of Incretin Analogs. A Preliminary Study
Brief Title: Stress Hyperglycemia. Potential Role of Incretin Analogs
Status: Completed | Type: Observational
Sponsor: Hospital Universitari Son Dureta (Other)
Collaborators: Fundació Mateu Orfila (Unknown)
Responsible Party: Juan A Llompart-Pou, Hospital Universitari Son Dureta
Other Study IDs: Incretins2010
Record Dates: First submitted 2010-03-11; First posted 2010-03-16 (Estimated); Last update posted 2010-06-08 (Estimated); Status verified 2010-06

CONDITIONS: Hyperglycemia; Critical Illness
Keywords: Stress hyperglycemia; Incretins; GLP-1; GIP; glucoregulatory hormones
MeSH Terms: conditions — Hyperglycemia; Critical Illness

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Plasma and serum samples to analyze glucorregulatory hormones.
Oversight: Data Monitoring Committee: No

SUMMARY:
This is a prospective observational study to examine the levels of glucoregulatory hormones, with special focus on incretins levels, in critically ill patients with stress hyperglycemia.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years
* Emergent ICU admission
* Written informed consent from patient or relative.

Exclusion Criteria:

* Previously known type I or type II diabetes.
* Patients who received insulin or oral antidiabetic agents before ICU admission.
* Malignancies.
* Scheduled surgery
* Patients receiving enteral or parenteral nutrition.
* Inability to obtain informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Medical-surgical ICU patients
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2010-01; Primary Completion 2010-04 (Actual); Study Completion 2010-04 (Actual)

PRIMARY OUTCOMES:
Incretins plasmatic levels | 28 days
  28 days and ICU mortality

SECONDARY OUTCOMES:
glucagon | 28 days
  28 days and ICU mortality
insulin | 28 days
  28 days and ICU mortality
cortisol | 28 days
  28 days and ICU mortality
HOMA index | 28 days
  28 days and ICU mortality

CONTACTS AND LOCATIONS:
Overall Officials: Juan A Llompart-Pou, M.D., Principal Investigator — Hospital Universitari Son Dureta. Intensive Care Unit
Locations (1):
- Hospital Universitari Son Dureta. Intensive Care Unit, Palma de Mallorca, Balearic Islands, Spain

REFERENCES:
- [Derived] Llompart-Pou JA, Fernandez-de-Castillo AG, Burguera B, Perez-Barcena J, Marse P, Rodriguez-Yago M, Barcelo A, Raurich JM. Stress hyperglycaemia in critically ill patients: potential role of incretin hormones; a preliminary study. Nutr Hosp. 2012 Jan-Feb;27(1):130-7. doi: 10.1590/S0212-16112012000100015. PMID 22566312